CLINICAL TRIAL: NCT04665323
Title: An International Cross-sectional Survey to Evaluate the Burden of Fibrodysplasia Ossificans Progressiva (FOP) on Patients and Their Families.
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-60120-450
Record Dates: First submitted 2020-11-25; First posted 2020-12-11 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Fibrodysplasia Ossificans Progressiva
MeSH Terms: conditions — Myositis Ossificans

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (4):
- People living with FOP
- Parent or legal guardian primary caregivers
- Parent or legal guardian
- Siblings

SUMMARY:
The FOP burden of illness (BoI) survey aims to assess the impact of the burden of FOP on patients and their families. The study is being conducted online and available for residents in Argentina, Brazil, Canada, France, Germany, Italy, Japan, Mexico, Poland, Russia, South Korea, Spain, Sweden, the US, and the UK.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals meeting one of the two categories below (A or B) are eligible to participate: A. Any individual with FOP, of any age; B. Any individual who is a family member of a person with FOP (i.e. either a parent / legal guardian or a sibling) and who is aged 18 years and older
2. All adult participants and parents / legal guardians of minors should provide informed consent before starting filling out the survey

Exclusion Criteria:

1. Any individuals who are unable to complete the online survey independently or to get assistance to physically enter the answers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Convenience Sample
Sampling Method: Non-Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Quality of life of people living with FOP and their family members, measured using the EuroQol health-related quality of life (QoL) questionnaire (EQ-5D-5L) | Baseline
Quality of life of people living with FOP and their family members, measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) | Baseline
Caregiver burden for the parent primary caregiver, measured using the Zarit Burden Interview (ZBI) | Baseline
Responses to bespoke questionnaire describing the emotional burden on family members | Baseline
Physical function of the person living with FOP, measured using the FOP Physical Function Questionnaire (FOP-PFQ). | Baseline
Joint function of the person living with FOP, measured using Patient-Reported Mobility Assessment (PRMA). | Baseline
Responses to bespoke questionnaire describing the types of healthcare services utilized by the person living with FOP over the last two years | Baseline
Responses to bespoke questionnaire describing the frequency of utilization of healthcare services by the person living with FOP over the last two years. | Baseline
Responses to bespoke questionnaire describing the impact of FOP on modifications to the living environment (e.g. home modifications) and travels. | Baseline
Responses to bespoke questionnaire describing the expenses paid by the family for the care of the person living with FOP | Baseline
Responses to bespoke questionnaire describing the Impact of FOP on education, employment, and career choices for people living with FOP and their family members | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Ipsen Central Contact, Cambridge, Massachusetts, United States